CLINICAL TRIAL: NCT07240350
Title: The Role and Regulatory Mechanism of Germinal Center Immune Response in Hepatitis B Virus Infection
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-279
Record Dates: First submitted 2025-06-19; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hepatitis B Virus Infection
Keywords: Germinal center; humoral immunity; immune response; hepatitis B virus infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBV patients who underwent liver, spleen, tonsil, and lymph node surgery: The group of HBV patients who underwent liver, spleen, tonsil, and lymph node surgery.
  Interventions: Procedure: Tissue resection
- Healthy patients who underwent liver, spleen, tonsil, and lymph node surgery: The group of HBV patients who underwent liver, spleen, tonsil, and lymph node surgery.
  Interventions: Procedure: Tissue resection

INTERVENTIONS:
Procedure: Tissue resection — The group of HBV patients who underwent liver, spleen, tonsil, and lymph node surgery and the group of HBV-negative patients who underwent liver, spleen, tonsil, and lymph node surgery

SUMMARY:
The purpose of this observational study is to investigate the structure and composition of germinal centers in individuals with chronic HBV infection. The primary questions it aims to address are:

What are the phenotypes, functions, and complexity of B cell clones of the immune cells within the germinal centers of chronic HBV-infected individuals? Do chronic HBV-infected individuals have ectopic germinal centers in the liver? This will be studied by collecting peripheral blood and discarded liver, lymph node, and tonsil tissues from chronic HBV patients undergoing lymph node surgery, hepatectomy, and tonsillectomy.

DETAILED DESCRIPTION:
This study is a single-center, prospective, cross-sectional investigation. We plan to enroll 280 participants.By collecting discarded liver, spleen, tonsil, and lymph node tissues from chronic HBV-infected and HBsAg-negative patients postoperatively, we aim to compare the phenotypic and functional differences of various immune cells in the germinal centers of these organs between the two groups. We will also identify the HBV antigen specificity of B cell clones in different germinal centers. Additionally, we will observe the structural, transcriptomic, and proteomic differences in germinal center tissues between the two groups to elucidate the impact of chronic HBV infection on germinal centers. During the study, no random or protocol-driven treatments will be administered to participants. If clinically appropriate, the treating physician will make decisions and select treatment plans based on individual circumstances.

Data Collection Procedures Since this is a single-center, prospective, cross-sectional study, no additional visits or laboratory analyses beyond routine clinical practice are required. Physicians will determine treatment plans in accordance with instructions and local guidelines. Researchers will review patients' medical histories and laboratory reports to determine eligibility based on inclusion and exclusion criteria. Patients must sign the most recent informed consent form (ICF) approved by the IRB/IEC before data collection. In line with routine clinical practice, surgeons will prioritize clinical needs when obtaining surgical specimens, and then collect discarded clinical samples for experimental exploration and clinical data analysis. Each participant will be assigned a unique identification number, such as HBV-liver/tonsil/LN/spleen-1, HBV-liver/tonsil/LN/spleen-2, HC-liver/tonsil/LN/spleen-1, HC-liver/tonsil/LN/spleen-2, etc. All study documents (e.g., case report forms, clinical records) will use this identification number. In compliance with data privacy regulations, the use of unique identification numbers is permitted as long as they do not contain combinations of information that could identify participants (for example, the use of participants' initials and date of birth together is not allowed).

Sample Collection Demographic Data Recording: Record date of birth, gender, and initials. Medical History and Physical Examination: Include vital signs, height, weight, physical examination of all body systems; past and present medical history, including the presence of spider angiomas or palmar erythema, dull complexion, jaundice of skin and sclera, hepatic pain, and enlargement of liver, spleen, or lymph nodes.

Preoperative Peripheral Blood Collection: Draw 30 milliliters of peripheral blood from the subject's upper limb before surgery.

Collection of Discarded Liver , Spleen ,Tonsil, Lymph Node Tissue During Surgery: From subjects undergoing hepatectomy, tonsillectomy, splenectomy, or lymph node dissection, collect discarded liver, spleen ,tonsil, lymph node tissue during the surgical procedure.

Safety Monitoring, Reporting, and Medical Management Adverse Event (AE) Definition: An adverse event is any unfavorable medical occurrence in a patient or subject after the administration of a drug, whether or not considered related to the treatment. Adverse events can include any adverse signs (including abnormal laboratory findings), symptoms, or diseases temporally related to the use of the study drug, regardless of whether a causal relationship with the study drug is considered. Adverse events include both serious adverse events (SAEs) and non-serious adverse events.

SAE Definition: An SAE is a medical event occurring during a clinical study that requires hospitalization or prolongation of hospital stay, results in disability, affects the ability to work, is life-threatening or fatal, or causes congenital anomalies. These medical events include:

Events leading to death; Life-threatening events (defined as events where the subject is at immediate risk of death at the time of the event); Events requiring hospitalization or prolongation of hospital stay; Events that may result in permanent or significant disability

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, patients with chronic hepatitis B and hepatitis B surface antigen negative patients with clinical diagnosis who need to undergo liver, spleen, tonsil or lymph node surgery.
2. Before performing any research-related steps, the patient understood the research process, signed the informed consent, and complied with the research requirements.
3. Patients diagnosed with chronic hepatitis B virus infection according to the "Guidelines for the Prevention and Treatment of Chronic Hepatitis B(2019 Version)" .

Exclusion Criteria:

1. Those concomitant HCV, HIV infection, alcoholic fatty liver disease, non-alcoholic fatty liver disease, and autoimmune liver disease , etc. were excluded.
2. Diseases of the immune system or coagulation system, such as hyperthyroidism, diabetes, thrombocytopenic purpura, etc., were excluded.
3. Exclude serious underlying diseases that affect the immune status of the body.
4. The investigator believes that there are other circumstances that are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The group of HBV patients who underwent liver, spleen, tonsil, and lymph node surgery and the group of HBV-negative patients who underwent liver, spleen, tonsil, and lymph node surgery
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
The HBV-specific immune response levels will be measured using the immune cells from lymphoid follicle of the enrolled patients | After the tissue section collected
  Tissue section from the enrolled patients will be used to detect the levels of HBV-specific immunity and other laboratory indicators after restimulation with HBV peptide pools.

SECONDARY OUTCOMES:
Germinal center organization structure, transcriptomics and proteomics will be measured using the tissue section of the enrolled patients | After the tissue section collected
  We will utilize tissue samples and employ experimental methods such as immunohistochemistry, immunofluorescence, and spatial transcriptomics to measure the structure and size of germinal centers.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Southern Medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No